CLINICAL TRIAL: NCT02988427
Title: Measuring Patient Engagement in Diabetes Care
Status: Withdrawn | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: University of North Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: STU00203715
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
We will develop a new measure of patient engagement/activation specific to the context of diabetes self-care

ELIGIBILITY:
Inclusion Criteria:

1. Patient is age 21 and older
2. Patient is English speaking
3. Patient has been diagnosed with Type II Diabetes by a health care provider

Exclusion Criteria:

1. Severe, uncorrectable vision
2. Hearing impairments
3. Cognitive impairment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients ages 21 and older will be recruited from study clinics
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-efficacy | Baseline
  Self-efficacy will be assessed using an 8-item measure developed by Sarkar and colleagues asking respondents to rate their confidence in their ability to perform individual diabetes self-care activities, such as monitoring their blood glucose, getting medical attention, and taking care of their health.

SECONDARY OUTCOMES:
Diabetes Distress | Baseline
  The Diabetes Distress Scale (DDS) is a 17-item measure of diabetes-related emotional distress. It has four subscales corresponding to emotional burden, physician-related distress, regimen distress, and diabetes interpersonal distress.
Functional Health Status | Baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) is a national resource providing state-of-the-art tools for assessing patient symptoms and health outcomes. Short form measures of physical health (function) and emotional health (depression, anxiety) will be collected.
Clinical Outcomes | 3 months before baseline to 3 months after baseline
  Hemoglobin A1c (HbA1c) and LDL cholesterol lab values, along with systolic and diastolic blood pressure values are collected as part of routine clinical care at every 3 months, and will be recorded from the medical record from the most recent visit.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolf, PhD, MPH, MA, Principal Investigator — Northwestern University; Stacy Bailey, PhD, MPH, Principal Investigator — University of North Carolina

IPD SHARING:
Plan to Share IPD: No